CLINICAL TRIAL: NCT04576702
Title: A Phase 2, Randomized, Stratified, Observer-Blind Clinical Study to Evaluate Safety and Immunogenicity of an MF59-Adjuvanted Quadrivalent Subunit Inactivated Influenza Vaccine in Older Adults
Brief Title: Safety and Immunogenicity of an MF59-Adjuvanted Influenza Vaccine in Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V200_10
Record Dates: First submitted 2020-09-17; First posted 2020-10-06 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Influenza; Human
Keywords: Influenza; Vaccine; MF59; Adjuvant
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Investigational aIIV4c group (Experimental): aIIV4c will be administered as a single dose intramuscularly on Day 1
  Interventions: Biological: Investigational aIIV4c
- licensed IIV4c group (Active Comparator): IIV4c will be administered as a single dose intramuscularly on Day 1
  Interventions: Biological: IIV4c
- licensed aIIV4 group (Active Comparator): aIIV4 will be administered as a single dose intramuscularly on Day 1
  Interventions: Biological: aIIV4
- licensed RIV4 group (Active Comparator): RIV4 will be administered as a single dose intramuscularly on Day 1
  Interventions: Biological: RIV4

INTERVENTIONS:
Biological: Investigational aIIV4c — Investigational MF59 Adjuvanted Cell-derived Quadrivalent Influenza vaccine, containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO (World Health Organization) for quadrivalent vaccines for the respective season.
  Arms: Investigational aIIV4c group
Biological: IIV4c — Licensed, Non-adjuvanted, Cell-derived Quadrivalent Influenza Vaccine containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO for quadrivalent vaccines for the respective season.
  Arms: licensed IIV4c group
Biological: aIIV4 — Licensed, MF59-Adjuvanted, egg-derived Quadrivalent Influenza Vaccine containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO for quadrivalent vaccines for the respective season.
  Arms: licensed aIIV4 group
Biological: RIV4 — Licensed, Recombinant Quadrivalent Influenza Vaccine containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO for quadrivalent vaccines for the respective season.
  Arms: licensed RIV4 group

SUMMARY:
This Phase 2, randomized, observer-blind, active controlled clinical study is evaluating the safety and immunogenicity of the investigational MF59-Adjuvanted Quadrivalent Subunit Inactivated Influenza Vaccine. Approximately 480 subjects are to be randomized into 1 of 4 possible treatment groups (investigational Influenza Vaccine or licensed Quadrivalent Influenza Vaccine comparators) at 120 participants per group. Every participant will receive an influenza vaccine injection on Day 1 and will be followed up for approximately 6 months following injection. The primary immunogenicity analysis is based on Day 29 serum.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals 50 years of age and older on the day of informed consent.
2. Individuals who have voluntarily given written consent after the nature of the study has been explained according to local regulatory requirements, prior to study entry.
3. Individuals who can comply with study procedures including follow-up.
4. Males, females of non-childbearing potential or females of childbearing potential who are using an effective birth control method, at least 30 days prior to informed consent, which they intend to use for at least 2 months after the study vaccination.

Exclusion Criteria:

1. Females of childbearing potential who are pregnant, lactating, or who have not adhered to a specified set of contraceptive methods from at least 30 days prior to informed consent and who do not plan to do so until 2 months after the study vaccination.
2. Progressive, unstable or uncontrolled clinical conditions.
3. Hypersensitivity, including allergy, to any component of vaccines, medicinal products or medical equipment whose use is foreseen in this study.
4. History of any medical condition considered an adverse event of special interest.
5. Known history of Guillain Barré syndrome or another demyelinating disease such as encephalomyelitis and transverse myelitis.
6. Clinical conditions representing a contraindication to intramuscular administration of vaccines or blood draw.
7. Abnormal function of the immune system resulting from:

   1. Clinical conditions
   2. Systemic administration of corticosteroids (PO/IV/IM) at a dose of ≥ 20 mg/day of prednisone or equivalent for more than 14 consecutive days within 90 days prior to informed consent5.
   3. Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to informed consent.
8. Received immunoglobulins or any blood products within 180 days prior to informed consent.
9. Received an investigational or non-registered medicinal product within 30 days prior to vaccination.
10. Individuals who received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrolment in this study or who are planning to receive any vaccine within 28 days from the study vaccines.
11. Study personnel or immediate family or household member of study personnel.
12. Receipt of any influenza vaccine within 6 months prior to vaccination in this study, or plan to receive an influenza vaccine during the study period.
13. Acute (severe) febrile illness
14. Any other clinical condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subject due to participation in the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Director, Study Director — Seqirus
Locations (21):
- United States (21):
  - 4022 - Coastal Clinical Research, an AMR company, Mobile, Alabama
  - 4002 - Clinical Research Consortium, an AMR company, Tempe, Arizona
  - 4006 - Westside Center for Clinical Research, Jacksonville, Florida
  - 4013 - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - 4021 - Research Centers of America, LLC, Oakland, Florida
  - 4023 - Advanced Clinical Research, Boise, Idaho
  - 4010 - Heartland Research Associates, LLC, Newton, Kansas
  - 4016 - Heartland Research Associates, LLC - An AMR Company, Wichita, Kansas
  - 4001 - Central Kentucky Research Associates, an AMR company, Lexington, Kentucky
  - 4014 - Medpharmi, Kenner, Louisiana
  - 4008 - The Center for Pharmaceutical Research, an AMR company, Kansas City, Missouri
  - 4024 - Sundance Clinical Research, LLC, St Louis, Missouri
  - 4009 - Meridian Clinical Research, LLC, Omaha, Nebraska
  - 4007 - Regional Clinical Research / United Medical Associates, Binghamton, New York
  - 4012 - M3 Wake Research, Inc., Raleigh, North Carolina
  - 4004 - Sterling research, Cincinnati, Ohio
  - 4017 - Rapid Medical Research, Inc., Cleveland, Ohio
  - 4011 - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - 4005 - Clinical Trials of Texas, Inc., San Antonio, Texas
  - 4018 - Martin Diagnostic Clinic, Tomball, Texas
  - 4020 - Advanced Clinical Research, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
SEQIRUS supports the release of anonymized subject-level and study-level data in compliance with regulatory requirements, including Clinical Documents which are part of the Common Technical Documents (CTD) modules submitted to regulatory agencies for public release.
  Summary results disclosure is either in document form (e.g., International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) E3 Clinical Study Report synopsis) or structured data form (such as summary results in ClinicalTrials.gov (United States) or eudract.ema.europa.eu (EU Clinical Trial Registry [EU CTR])
Supporting Information: Study Protocol, SAP
Time Frame: SEQIRUS discloses results from clinical studies within 12 months of last patient last visit (LPLV) unless otherwise mandated by local laws or regulations.
Access Criteria: SEQIRUS will consider requests from qualified scientific and medical researchers to disclose protocols, anonymized subject-level data and study-level data when there is medical, scientific and/or public health interest to ensure the safe use of a Seqirus product licensed on or after 1 January 2014 in the United States (US) and/or the European Union (EU). This applies to Seqirus-sponsored interventional studies initiated after 27 September 2007 and ongoing as of 26 December 2007, that have been included as part of a US or EU submission package which received approval in US and EU on or after 1 January 2014 and have been accepted for publication
URL: http://ClinicalTrials.gov

REFERENCES:
- [Derived] Essink BJ, Vermeulen W, Andrade C, de Rooij R, Isakov L, Casula D, Albano FR. A randomised phase 2 immunogenicity and safety study of a MF59-adjuvanted quadrivalent subunit inactivated cell-derived influenza vaccine (aQIVc) in adults aged 50 years and older. Vaccine. 2025 Apr 2;51:126791. doi: 10.1016/j.vaccine.2025.126791. Epub 2025 Feb 12. PMID 39946829

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational aIIV4c Group | Licensed IIV4c Group | Licensed aIIV4 Group | Licensed RIV4 Group
Started | 116 | 119 | 116 | 120
Completed | 112 | 114 | 112 | 116
Not Completed | 4 | 5 | 4 | 4
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 3 | 3 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational aIIV4c Group | Licensed IIV4c Group | Licensed aIIV4 Group | Licensed RIV4 Group | Total
Number analyzed (Participants) | 116 | 119 | 116 | 120 | 471
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 56 | 57 | 56 | 58 | 227
  >=65 years | 60 | 62 | 60 | 62 | 244
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (9.18) | 64.7 (8.49) | 65.0 (7.49) | 65.4 (9.02) | 65.0 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 72 | 71 | 71 | 283
  Male | 47 | 47 | 45 | 49 | 188
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 89 | 100 | 99 | 105 | 393
  Black or African American | 23 | 15 | 14 | 15 | 67
  Asian | 1 | 2 | 1 | 0 | 4
  American Indian or Alaska Native | 2 | 2 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Other | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 116 | 119 | 116 | 120 | 471
vaccinated within 3 previous influenza seasons [Count of Participants; unit: Participants]
  yes | 84 | 85 | 84 | 85 | 338
  no | 32 | 34 | 32 | 35 | 133

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity Endpoint: Geometric Mean Titer (GMT) Against the A/H1N1, B/Victoria and B/Yamagata Vaccine Strains by Hemagglutination Inhibition (HI) Assay and Against A/H3N2 Strain Using Microneutralization Assay Using Cell-derived Target Viruses
Time Frame: 28 days post-vaccination
Population: Per Protocol Set (PPS): All subjects in the Full Analysis Set (FAS) Immunogenicity who:
  * Correctly received the vaccine (ie, received the vaccine to which the subject was randomized).
  * Had no clinical study report (CSR)-reportable protocol deviation (PD) leading to exclusion (ie, impacting the results) as defined prior to unblinding.
  * Had immunogenicity assessments within the window of +/- 7 days around the Day 29 visit, and Day 1 sample taken within 3 days before vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Investigational aIIV4c Group | Licensed IIV4c Group | Licensed aIIV4 Group | Licensed RIV4 Group
Number analyzed (Participants) | 110 | 114 | 109 | 116
titer
  A/H1N1 Day 1 HI GMT | 19.5 [15.5 to 24.5] | 17.04 [13.6 to 21.3] | 21.85 [17.4 to 27.5] | 18.05 [14.5 to 22.5]
  A/H1N1 Day 29 HI GMT | 146.05 [116.1 to 183.7] | 111.38 [88.8 to 139.7] | 119.54 [95.0 to 150.5] | 173.08 [138.5 to 216.4]
  B/Yamagata Day 1 HI GMT | 16.95 [14.3 to 20.1] | 16.02 [13.5 to 19.0] | 14.59 [12.3 to 17.3] | 15.99 [13.5 to 18.9]
  B/Yamagata Day 29 HI GMT | 69.35 [58.7 to 81.9] | 50.99 [43.3 to 60.1] | 37.51 [31.7 to 44.4] | 60.25 [51.2 to 70.8]
  B/Victoria Day 1 HI GMT | 21.86 [18.5 to 25.8] | 22.02 [18.7 to 25.9] | 20.42 [17.3 to 24.2] | 24.82 [21.1 to 29.2]
  B/Victoria Day 29 HI GMT | 94.82 [80.4 to 111.8] | 69.49 [59.1 to 81.7] | 52.35 [44.3 to 61.8] | 75.50 [64.3 to 88.6]
  A/H3N2 Day 1 MN GMT | 71.44 [61.7 to 82.7] | 59.37 [51.4 to 68.6] | 60.20 [52.0 to 69.7] | 64.93 [56.3 to 74.9]
  A/H3N2 Day 29 MN GMT | 138.88 [120.7 to 159.8] | 117.28 [102.2 to 134.6] | 106.22 [92.3 to 122.3] | 174.78 [152.6 to 200.2]

2. Primary Outcome: Immunogenicity Endpoint: Geometric Mean Ratio (GMR) (GMR is GMT Ratio of aIIV4c/Comparator) Against the A/H1N1, B/Victoria and B/Yamagata Vaccine Strains by HI Assay and Against A/H3N2 Strain Using MN Assay Using Cell-derived Target Viruses
Time Frame: 28 days post-vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Licensed IIV4c Group | Licensed aIIV4 Group | Licensed RIV4 Group
Number analyzed (Participants) | 114 | 109 | 116
Ratio
  A/H1N1 HI GMR (aIIV4c/comparator group) | 1.31 [0.96 to 1.79] | 1.22 [0.89 to 1.68] | 0.84 [0.62 to 1.15]
  B/Yamagata HI GMR (aIIV4c/comparator group) | 1.36 [1.08 to 1.71] | 1.85 [1.47 to 2.33] | 1.15 [0.92 to 1.44]
  B/Victoria HI GMR (aIIV4c/comparator group) | 1.36 [1.09 to 1.71] | 1.81 [1.44 to 2.27] | 1.26 [1.00 to 1.57]
  A/H3N2 MN GMR (aIIV4c/comparator group) | 1.18 [0.98 to 1.43] | 1.31 [1.08 to 1.59] | 0.79 [0.66 to 0.96]

3. Primary Outcome: Immunogenicity Endpoint: Percentage of Subjects Achieving Seroconversion for the A/H1N1, B/Victoria and B/Yamagata Strains by HI Assay and Against A/H3N2 Strain Using MN Assay Using Cell-derived Target Viruses
Description: Seroconversion is defined as ≥4-fold increase in titer postvaccination in those with pre-vaccination titer above or equal to the Lower Limit of Quantitation (LLOQ) (≥1:10), or a post-vaccination titer ≥1:40 for subjects with baseline titer below the LLOQ (1:10) for HI titers
Time Frame: 28 days post-vaccination
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Investigational aIIV4c Group | Licensed IIV4c Group | Licensed aIIV4 Group | Licensed RIV4 Group
Number analyzed (Participants) | 110 | 114 | 109 | 116
percentage of subjects
  A/H1N1 HI seroconversion Day 29 | 61.8 [52.1 to 70.9] | 54.4 [44.8 to 63.7] | 50.5 [40.7 to 60.2] | 61.2 [51.7 to 70.1]
  B/Yamagata HI seroconversion Day 29 | 42.7 [33.3 to 52.5] | 31.6 [23.2 to 40.9] | 19.3 [12.3 to 27.9] | 37.9 [29.1 to 47.4]
  B/Victoria HI seroconversion Day 29 | 46.4 [36.8 to 56.1] | 33.3 [24.8 to 42.8] | 26.6 [18.6 to 35.9] | 40.5 [31.5 to 50.0]
  A/H3N2 MN seroconversion Day 29 | 21.8 [14.5 to 30.7] | 20.2 [13.2 to 28.7] | 9.2 [4.5 to 16.2] | 32.8 [24.3 to 42.1]

4. Primary Outcome: Immunogenicity Endpoint: Percentage of Subjects With HI Titer ≥1:40 for A/H1N1, B/Yamagata and B/Victoria Strains (HI Assay) Using Cell-derived Target Viruses
Time Frame: 28 days post-vaccination
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Investigational aIIV4c Group | Licensed IIV4c Group | Licensed aIIV4 Group | Licensed RIV4 Group
Number analyzed (Participants) | 110 | 114 | 109 | 116
percentage of subjects
  A/H1N1 Day 1 | 44.5 [35.1 to 54.3] | 36.8 [28.0 to 46.4] | 41.3 [31.9 to 51.1] | 38.8 [29.9 to 48.3]
  A/H1N1 Day 29 | 85.5 [77.5 to 91.5] | 81.6 [73.2 to 88.2] | 82.6 [74.1 to 89.2] | 84.5 [76.6 to 90.5]
  B/Yamagata day 1 | 27.3 [19.2 to 36.6] | 23.7 [16.2 to 32.6] | 20.2 [13.1 to 28.9] | 28.4 [20.5 to 37.6]
  B/Yamagata Day 29 | 81.8 [73.3 to 88.5] | 64.0 [54.5 to 72.8] | 52.3 [42.5 to 61.9] | 65.5 [56.1 to 74.1]
  B/Victoria Day 1 | 32.7 [24.1 to 42.3] | 32.5 [24.0 to 41.9] | 30.3 [21.8 to 39.8] | 38.8 [29.9 to 48.3]
  B/Victoria Day 29 | 90.0 [82.8 to 94.9] | 72.8 [63.7 to 80.7] | 69.7 [60.9 to 78.2] | 79.3 [70.8 to 86.3]

5. Secondary Outcome: Safety Endpoint: The Percentage of Subjects With Solicited Local and Systemic Reactions
Description: The percentage of subjects with at least one solicited AE Day 1 through Day 7 after study vaccination.
Time Frame: 7 days post-vaccination
Population: Solicited Safety Set, defined as all subjects in the FAS with any solicited AE data.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational aIIV4c Group | Licensed IIV4c Group | Licensed aIIV4 Group | Licensed RIV4 Group
Number analyzed (Participants) | 115 | 117 | 114 | 119
Participants
  solicited AEs | 85 | 72 | 83 | 80
  Solicited local AEs | 70 | 52 | 67 | 51
  Solicited systemic AEs | 69 | 51 | 57 | 64
  analgesic/antipyretic use | 18 | 9 | 11 | 9

6. Secondary Outcome: Safety Endpoint: The Percentage of Subjects With Any Unsolicited Adverse Events
Description: The percentage of subjects with at least one unsolicited AE from Day 1 to Day 29.
  Related AEs = considered at least possibly related to study vaccination by the investigator.
Time Frame: 28 days post-vaccination
Population: Unsolicited Safety Set, defined as all subjects in the FAS with any unsolicited AE data
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational aIIV4c Group | Licensed IIV4c Group | Licensed aIIV4 Group | Licensed RIV4 Group
Number analyzed (Participants) | 116 | 119 | 116 | 120
Participants
  Any Unsolicited AE | 23 | 27 | 23 | 29
  Any Related Unsolicited AE | 1 | 1 | 3 | 0

7. Secondary Outcome: Safety Endpoint: The Percentage of Subjects With Serious Adverse Events (SAEs), AEs Leading to Withdrawal, Adverse Events of Special Interest (AESI) and Medically Attended Adverse Events (MAAEs) During the Entire Study Period
Time Frame: 180 days post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational aIIV4c Group | Licensed IIV4c Group | Licensed aIIV4 Group | Licensed RIV4 Group
Number analyzed (Participants) | 116 | 119 | 116 | 120
Participants
  Any Serious Unsolicited AE | 2 | 1 | 4 | 6
  Any Related Serious Unsolicited AE | 0 | 0 | 0 | 0
  Any Unsolicited AE of Special Interest | 1 | 0 | 0 | 0
  Any Medically Attended AE | 21 | 13 | 15 | 21
  Any Unsolicited AE Leading to Withdrawal from the Study | 1 | 0 | 0 | 0
  Any Death | 1 | 0 | 0 | 0

8. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Titer (GMT) Against the A/H1N1, B/Victoria and B/Yamagata Vaccine Strains by Microneutralization (MN) Assay Using Cell-derived Target Viruses
Time Frame: 28 days post-vaccination
Population: Per Protocol Set (PPS): All subjects in the FAS Immunogenicity who:
  * Correctly received the vaccine (ie, received the vaccine to which the subject was randomized).
  * Had no CSR-reportable PD leading to exclusion (ie, impacting the results) as defined prior to unblinding.
  * Had immunogenicity assessments within the window of +/- 7 days around the Day 29 visit, and Day 1 sample taken within 3 days before vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Investigational aIIV4c Group | Licensed IIV4c Group | Licensed aIIV4 Group | Licensed RIV4 Group
Number analyzed (Participants) | 110 | 114 | 109 | 116
titer
  A/H1N1 Day 1 | 158.64 [122.0 to 206.3] | 102.88 [79.5 to 133.1] | 162.19 [124.6 to 211.1] | 138.73 [107.5 to 179.0]
  A/H1N1 Day 29 | 1261.77 [997.2 to 1596.5] | 1036.72 [820.3 to 1310.3] | 1050.54 [829.5 to 1330.4] | 1719.68 [1368.0 to 2161.7]
  B/Yamagata Day 1 | 19.48 [17.0 to 22.3] | 15.55 [13.6 to 17.8] | 17.50 [15.2 to 20.1] | 17.62 [15.4 to 20.1]
  B/Yamagata Day 29 | 48.08 [41.9 to 55.2] | 42.89 [37.4 to 49.1] | 39.01 [34.0 to 44.8] | 56.12 [49.1 to 64.1]
  B/Victoria Day 1 | 18.63 [16.1 to 21.6] | 15.71 [13.6 to 18.1] | 18.02 [15.6 to 20.9] | 18.02 [15.7 to 20.8]
  B/Victoria Day 29 | 58.47 [50.4 to 67.8] | 47.63 [41.1 to 55.2] | 44.88 [38.7 to 52.1] | 61.8 [53.5 to 71.4]

9. Secondary Outcome: Immunogenicity Endpoint: GMR (GMR is GMT Ratio of aIIV4c/Comparator) Against the A/H1N1, B/Victoria and B/Yamagata Vaccine Strains by Microneutralization Assay Using Cell-derived Target Viruses
Time Frame: 28 days post-vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Licensed IIV4c Group | Licensed aIIV4 Group | Licensed RIV4 Group
Number analyzed (Participants) | 114 | 109 | 116
ratio
  A/H1N1 Day 29 MN GMR (aIIV4c/comparator group) | 1.22 [0.88 to 1.68] | 1.20 [0.87 to 1.66] | 0.73 [0.53 to 1.01]
  B/Yamagata Day 29 MN GMR (aIIV4c/comparator group) | 1.12 [0.93 to 1.35] | 1.23 [1.02 to 1.49] | 0.86 [0.71 to 1.03]
  B/Victoria Day 29 MN GMR (aIIV4c/comparator group) | 1.23 [1.00 to 1.50] | 1.30 [1.06 to 1.60] | 0.95 [0.77 to 1.16]

10. Secondary Outcome: Immunogenicity Endpoint: Percentage of Subjects Achieving Seroconversion for the A/H1N1, B/Victoria and B/Yamagata Strains by MN Assay Using Cell-derived Target Viruses
Description: as for outcome 3
Time Frame: 28 days post-vaccination
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Investigational aIIV4c Group | Licensed IIV4c Group | Licensed aIIV4 Group | Licensed RIV4 Group
Number analyzed (Participants) | 110 | 114 | 109 | 116
percentage of subjects
  A/H1N1 Day 29 | 61.8 [52.1 to 70.9] | 60.5 [50.9 to 69.6] | 53.2 [43.4 to 62.8] | 70.7 [61.5 to 78.8]
  B/Yamagata Day 29 | 22.7 [15.3 to 31.7] | 28.1 [20.1 to 37.3] | 15.6 [9.4 to 23.8] | 33.6 [25.1 to 43.0]
  B/Victoria Day 29 | 29.1 [20.8 to 38.5] | 26.3 [18.5 to 35.4] | 22.0 [14.6 to 31.0] | 37.1 [28.3 to 46.5]

11. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Titer (GMT) Against the A/H1N1, B/Victoria and B/Yamagata Vaccine Strains by Hemagglutination Inhibition (HI) Assay Using Cell-derived Target Viruses
Time Frame: 180 days post-vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Investigational aIIV4c Group | Licensed IIV4c Group | Licensed aIIV4 Group | Licensed RIV4 Group
Number analyzed (Participants) | 108 | 110 | 110 | 113
titer
  A/H1N1 Day 181 | 156.47 [127.6 to 191.9] | 144.08 [117.6 to 176.5] | 157.72 [128.9 to 193.0] | 198.17 [162.3 to 242.0]
  B/Yamagata Day 181 | 34.70 [29.2 to 41.3] | 33.26 [28.0 to 39.5] | 23.56 [19.8 to 28.0] | 32.04 [27.0 to 38.0]
  B/Victoria Day 181 | 103.64 [88.6 to 121.3] | 94.16 [80.6 to 110.0] | 67.78 [58.0 to 79.2] | 74.54 [63.9 to 86.9]

12. Secondary Outcome: Immunogenicity Endpoint: GMR (GMR is GMT Ratio of aIIV4c/Comparator) Against the A/H1N1, B/Victoria and B/Yamagata Vaccine Strains by Hemagglutination Inhibition (HI) Assay Using Cell-derived Target Viruses
Time Frame: 180 days post-vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Licensed IIV4c Group | Licensed aIIV4 Group | Licensed RIV4 Group
Number analyzed (Participants) | 110 | 110 | 113
Ratio
  A/H1N1 Day 181 HI GMR (aIIV4c/comparator group) | 1.09 [0.82 to 1.44] | 0.99 [0.75 to 1.31] | 0.79 [0.60 to 1.04]
  B/Yamagata Day 181 HI GMR (aIIV4c/comparator group) | 1.04 [0.82 to 1.32] | 1.47 [1.16 to 1.87] | 1.08 [0.86 to 1.37]
  B/Victoria Day 181 HI GMR (aIIV4c/comparator group) | 1.10 [0.89 to 1.36] | 1.53 [1.23 to 1.90] | 1.39 [1.12 to 1.72]

13. Secondary Outcome: Immunogenicity Endpoint: Percentage of Subjects With HI Titer ≥1:40 for A/H1N1, B/Yamagata and B/Victoria Strains (HI Assay) Using Cell-derived Target Viruses
Time Frame: 180 days post-vaccination
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Investigational aIIV4c Group | Licensed IIV4c Group | Licensed aIIV4 Group | Licensed RIV4 Group
Number analyzed (Participants) | 108 | 110 | 110 | 113
percentage of subjects
  A/H1N1 Day 181 | 88.9 [81.4 to 94.1] | 87.3 [79.6 to 92.9] | 87.3 [79.6 to 92.9] | 87.6 [80.1 to 93.1]
  B/Yamagata Day 181 | 50.0 [40.2 to 59.8] | 50.0 [40.3 to 59.7] | 32.7 [24.1 to 42.3] | 52.2 [42.6 to 61.7]
  B/Victoria Day 181 | 93.5 [87.1 to 97.4] | 91.8 [85.0 to 96.2] | 77.3 [68.3 to 84.7] | 82.3 [74.0 to 88.8]

14. Secondary Outcome: Immunogenicity Endpoint: Geometric Mean Titer (GMT) Against the A/H1N1, A/H3N2, B/Victoria and B/Yamagata Vaccine Strains by MN Assay Using Cell-derived Target Viruses
Time Frame: 180 days post-vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Investigational aIIV4c Group | Licensed IIV4c Group | Licensed aIIV4 Group | Licensed RIV4 Group
Number analyzed (Participants) | 108 | 110 | 110 | 113
titer
  A/H1N1 Day 181 | 481.49 [378.4 to 612.6] | 523.03 [410.7 to 666.0] | 502.85 [396.2 to 638.2] | 841.31 [664.8 to 1064.7]
  A/H3N2 Day 181 | 68.72 [56.9 to 83.1] | 68.17 [56.5 to 82.3] | 54.35 [45.0 to 65.6] | 100.14 [83.2 to 120.5]
  B/Yamagata Day 181 | 24.46 [21.5 to 27.8] | 24.98 [22.0 to 28.4] | 21.82 [19.2 to 24.8] | 28.17 [24.8 to 32.0]
  B/Victoria Day 181 | 31.68 [27.4 to 36.7] | 27.39 [23.7 to 31.7] | 24.97 [21.6 to 28.9] | 34.09 [29.5 to 39.3]

15. Secondary Outcome: Immunogenicity Endpoint: GMR (GMR is GMT Ratio of aIIV4c/Comparator) Against the A/H1N1, A/H3N2, B/Victoria and B/Yamagata Vaccine Strains by MN Assay Using Cell-derived Target Viruses
Time Frame: 180 days post-vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Licensed IIV4c Group | Licensed aIIV4 Group | Licensed RIV4 Group
Number analyzed (Participants) | 110 | 110 | 113
ratio
  A/H1N1 day 181 MN GMR (aIIV4c/comparator group) | 0.92 [0.66 to 1.28] | 0.96 [0.69 to 1.33] | 0.57 [0.41 to 0.79]
  A/H3N2 Day 181 MN GMR (aIIV4c/comparator group) | 1.01 [0.78 to 1.31] | 1.26 [0.98 to 1.64] | 0.69 [0.53 to 0.89]
  B/Yamagata Day 181 MN GMR (aIIV4c/comparator group) | 0.98 [0.82 to 1.17] | 1.12 [0.94 to 1.34] | 0.87 [0.73 to 1.03]
  B/Victoria Day 181 MN GMR (aIIV4c/comparator group) | 1.16 [0.95 to 1.41] | 1.27 [1.04 to 1.55] | 0.93 [0.76 to 1.13]

ADVERSE EVENTS:
Time Frame: Time frame for all-cause mortality: 6 months SAEs: Day 1 to Day 181; Nonserious unsolicited AEs: Day 1 to Day 29; Solicited AEs: Day 1 to Day 7 after vaccination
Description: SAEs, nonserious unsolicited AEs, and solicited AEs are reported in this Adverse Events section.
Arm/Group | Investigational aIIV4c Group | Licensed IIV4c Group | Licensed aIIV4 Group | Licensed RIV4 Group
All-Cause Mortality (participants affected / at risk) | 1/116 | 0/119 | 0/116 | 0/120
Serious Adverse Events (participants affected / at risk) | 2/116 | 1/119 | 4/116 | 6/120
Other Adverse Events (participants affected / at risk) | 86/116 | 77/119 | 84/116 | 83/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Investigational aIIV4c Group (N=116) | Licensed IIV4c Group (N=119) | Licensed aIIV4 Group (N=116) | Licensed RIV4 Group (N=120)
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 1 | 2
Scrotal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational aIIV4c Group (N=116) | Licensed IIV4c Group (N=119) | Licensed aIIV4 Group (N=116) | Licensed RIV4 Group (N=120)
Nausea (Gastrointestinal disorders) | 16 (16) | 12 (12) | 13 (13) | 15 (15)
chills (General disorders) | 15 (15) | 8 (8) | 12 (12) | 12 (12)
fatigue (General disorders) | 50 (50) | 29 (29) | 30 (30) | 40 (40)
Induration (General disorders) | 6 (6) | 5 (5) | 6 (6) | 4 (4)
Injection site pain (General disorders) | 70 (70) | 51 (51) | 66 (66) | 51 (51)
loss of appetite (Metabolism and nutrition disorders) | 17 (17) | 13 (13) | 15 (15) | 20 (20)
arthralgia (Musculoskeletal and connective tissue disorders) | 35 (35) | 19 (19) | 23 (23) | 28 (28)
myalgia (Musculoskeletal and connective tissue disorders) | 40 (40) | 23 (23) | 26 (26) | 27 (27)
headache (Nervous system disorders) | 37 (37) | 28 (28) | 29 (29) | 36 (36)
erythema (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT04576702/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT04576702/SAP_001.pdf